CLINICAL TRIAL: NCT03034720
Title: Collaborative Care Model for the Treatment of Persistent Symptoms After Concussion Among Youth
Status: Completed | Phase: Not Applicable | Type: Interventional
Sponsor: Seattle Children's Hospital (Other)
Responsible Party: Principal Investigator, Fred Rivara, Investigator, Seattle Children's Hospital
Allocation: Randomized | Model: Parallel | Masking: Single | Purpose: Treatment
Other Study IDs: STUDY00000437
Record Dates: First submitted 2017-01-11; First posted 2017-01-27 (Estimated); Last update posted 2021-04-08 (Actual); Status verified 2021-04

CONDITIONS: Concussion, Brain; TBI; Depression; Anxiety
Keywords: Concussion; persistent post-concussive symptoms; CBT; collaborative care; Depression; Anxiety
MeSH Terms: conditions — Brain Concussion; Depression; Anxiety Disorders

STUDY DESIGN:
Who Masked: Outcomes Assessor
Oversight: Data Monitoring Committee: Yes | FDA-regulated Drug: No | FDA-regulated Device: No

ARMS (2):
- Intervention (Experimental): Intervention subjects will receive treatment from an MSW-trained care manager over the course of 6-months after randomization. Intervention team members will work collaboratively with primary care providers to link physical and mental health care longitudinally through outpatient follow-up and community rehabilitation. Intervention subjects and their families and collaborative team members will share information and deliberate treatment decisions with each other in order to develop an individually tailored treatment plan. Stepped, higher intensity care will be available for intervention subjects with recurrent symptoms. Stepped up care will include CBT booster sessions targeting post-concussive and related symptom comorbidity as well as psychopharmacologic assessment and treatment.
  Interventions: Behavioral: Collaborative Care
- Control (No Intervention): Adolescent subjects in the control group will receive care as usual from their health care providers, a standard that is ethically acceptable.

INTERVENTIONS:
Behavioral: Collaborative Care — Intervention subjects will receive treatment from an MSW-trained care manager over the course of 6-months after randomization. Intervention team members will work collaboratively with primary care providers to link physical and mental health care longitudinally through outpatient follow-up and community rehabilitation. Intervention subjects and their families and collaborative team members will share information and deliberate treatment decisions with each other in order to develop an individually tailored treatment plan. Stepped, higher intensity care will be available for intervention subjects with recurrent symptoms. Stepped up care will include CBT booster sessions targeting post-concussive and related symptom comorbidity as well as psychopharmacologic assessment and treatment.
  Arms: Intervention

SUMMARY:
SPECIFIC AIMS

While post-concussive symptoms following sports-related concussion are typically transient and resolve spontaneously within two weeks of concussive injury, 14% or more of youth who sustain concussion experience significant morbidity that can persist well beyond the normal disease course.Furthermore, post-concussive symptoms commonly co-occur with affective symptoms including depression and anxiety which when present can prolong recovery from primary post-concussive symptoms. Together, persistent physical and psychological symptoms confer protracted functional impairment and create a significant burden for affected youth, their family, and school. Currently, there are no evidence-based guidelines to inform treatment of persistent post-concussive symptoms in youth and adolescents.

In response to the dearth of evidence-based treatment approaches for youth with persistent post-concussive symptoms, the investigators developed a novel collaborative care treatment model that simultaneously targets post-concussive symptoms and co-occurring depression and anxiety. Athletes and their family members receive patient navigator care management services that bridge post-injury care across acute care, specialist and primary care health service delivery sectors, in addition to cognitive behavioral psychotherapy. Patients who remain symptomatic after initial treatment efforts receive stepped-up care that may include psychopharmacologic consultation. The Investigators have demonstrated feasibility of the intervention model through a pilot randomized-control trial of 49 adolescents with persistent post-concussive symptoms recruited from a regional children's hospital. Participants assigned to the intervention condition demonstrated significant and clinically-meaningful reductions in post-concussive and depressive symptoms as well as health-related quality of life as compared to adolescents in the usual care arm of the trial.

DETAILED DESCRIPTION:
The proposed study will expand upon the pilot trial in order to further develop, implement, and test the impact of an innovative collaborative care approach tailored to the needs of a patient population who currently have no evidence-based options. The investigators propose a broad reach intervention strategy that is designed to be readily implemented in acute, specialty and primary care medical settings, as well as over the telephone. The investigators will conduct a randomized comparative effectiveness trial with 200 youth, ages 11-18, suffering from ≥ 3 post-concussive symptoms at least 1 month after their sports-related injury. Athletes will be randomized to collaborative care (intervention) or post-sports injury care as usual (control group) conditions. The study is designed with the following aims:

Aim 1. To determine the effectiveness of a stepped-collaborative care intervention model in reducing post-concussive and co-occurring psychological symptoms in youth with persistent post-concussive symptoms after sports-related concussion H1: Youth receiving a collaborative care intervention will demonstrate clinically and statistically significant reductions in post-concussive symptoms, depressive and anxiety symptoms over the course of the 12-month study, compared to usual care control group athletes Aim 2. To examine the effectiveness of the intervention in improving function and health-related quality of life amongst youth with persistent symptoms after sports-related concussion H2: Adolescents who receive a collaborative care intervention will exhibit a clinically meaningful improvement in function and health-related quality life Exploratory Aim 3. To explore differences in school performance between groups H3: Adolescents who receive the collaborative care intervention will receive individualized treatment and community resource linkages which will improve their school performance as compared to adolescents receiving treatment as usual Aim 4. To explore the heterogeneity of treatment effects in the primary and secondary outcomes by examining the interaction of the treatment effect with group membership in distinct subgroups of the population. H4: Three distinct subgroups are expected to emerge from the study population: adolescents who recover from symptoms, adolescents with chronic psychosocial problems, and adolescents whose symptoms wax and wane over time. A greater proportion of adolescents who recover from symptoms will emerge in the treatment group, compared to controls.

IMPACT: By broadly targeting the constellation of post-concussive physical and psychological symptoms and integrating care amongst primary care, pediatric sub-specialist, and behavioral health providers, the collaborative care health services intervention could accelerate the rate of recovery from persistent post-concussive symptoms and attenuate the degree and duration of disability during adolescence, a critical period for healthy development. Validation of this treatment through a scaled up clinical trial will serve as a foundation for broader dissemination of this collaborative care treatment model. The multidisciplinary sports concussion research team will simultaneously work nationally and internationally to ensure study results are expediently translated into effective policy for youth athletes suffering from enduring symptoms and functional impairments in the wake of sports-related concussions.

ELIGIBILITY:
Inclusion Criteria:

* English speaking male and female sports-injured adolescents
* ages 11-18
* health care provider diagnosed concussion and with ≥ 3 HBI symptoms that have endured or worsened for at least 1-month but less than 9 months since injury will be included in the investigation.

Exclusion Criteria:

* Adolescents who require immediate intervention (e.g., acute suicidal ideation) will be excluded.
* Adolescents whose parents report that their child has ever had a diagnosis of schizophrenia or psychosis will be excluded from the study.
* Adolescents whose parents report concerns about their child's ability to communicate may be excluded from the study (pending consult with PIs).
* Adolescents who have suffered spinal cord or other severe injuries that prevent participation will be excluded from the study.

  * Adults unable to consent are not included in this research
  * Adolescents and parents who do not read and speak English will not be included
  * Wards of the state are not included in this research
  * Pregnant women are not included in this research
  * Prisoners are not included in this research

Ages: 11 Years to 18 Years | Sex: All | Healthy Volunteers: No
Age Groups: Child, Adult
Enrollment: 200 (Actual)
Dates: Start 2017-03-09 (Actual); Primary Completion 2020-05-29 (Actual); Study Completion 2020-05-29 (Actual)

PRIMARY OUTCOMES:
Post-concussive symptoms measured with the HBI | During the12 months after enrollment.
  The central hypothesis is that the two groups will have different patterns of HBI scores over time, with the intervention group showing significant. reductions when compared to controls.
Health related quality of life as measured with the PedsQL | During the 12 months after enrollment
  The hypothesis is that the two groups will have different patterns of PEDSQL scores over time, with the intervention group showing significant reductions when compared to controls.
Depressive symptoms measured by the PHQ-9 | During the12 months after enrollment.
  The hypothesis is that the two groups will have different patterns of PHQ-9 scores over time, with the intervention group showing significant. reductions when compared to controls.
Anxiety symptoms measured by the GAD-7 | During the 12 months after enrollment
  The hypothesis is that the two groups will have different patterns of GAD-7 scores over time, with the intervention group showing significant reductions when compared to controls.
Anxiety symptoms measured by the RCADS | During the 12 months after enrollment
  The hypothesis is that the two groups will have different patterns of RCADS scores over time, with the intervention group showing significant reductions when compared to controls.

SECONDARY OUTCOMES:
School performance as measured by GPA | During the 12 months after enrollment
Return to full activities at school as measured by the CLASS | During the 12 months after enrollment
  The secondary hypothesis is that the two groups will have different patterns on the CLASS over time, with the intervention group showing significant reductions when compared to controls

OTHER OUTCOMES:
Exploratory Outcome Measure | During the 12 months after enrollment
  Exploratory outcome measures: Heterogeneity of treatment effects in the primary and secondary outcomes by examining interaction between treatment group and membership in distinct subgroups of the study population representing youth who recover from symptoms, youth with chronic psychosocial problems, and youth whose symptoms wax and wane over follow up.

CONTACTS AND LOCATIONS:
Overall Officials: Frederick P Rivara, MD, Principal Investigator — Seattle Children's Hospital
Locations (1):
- Seattle Childrens Hospital, Seattle, Washington, United States

REFERENCES:
- [Background] Payne KM, Prentice ET, Marcynyszyn LA, McCarty CA. Goals for Persistent Postconcussive Symptom Treatment From Adolescent and Parent Perspectives. JAMA Pediatr. 2020 Dec 1;174(12):1210-1211. doi: 10.1001/jamapediatrics.2020.0898. PMID 32391873
- [Background] Marcynyszyn LA, McCarty CA, Rivara FP, Johnson AM, Wang J, Zatzick DF. Parent Traumatic Events and Adolescent Internalizing Symptoms: The Mediating Role of Parental Depression Among Youth with Persistent Post-concussive Symptoms. J Pediatr Psychol. 2021 Jun 3;46(5):547-556. doi: 10.1093/jpepsy/jsaa128. PMID 33411915
- [Background] McCarty CA, Zatzick D, Hoopes T, Payne K, Parrish R, Rivara FP. Collaborative care model for treatment of persistent symptoms after concussion among youth (CARE4PCS-II): Study protocol for a randomized, controlled trial. Trials. 2019 Sep 18;20(1):567. doi: 10.1186/s13063-019-3662-3. PMID 31533799
- [Background] Johnson AM, McCarty CA, Marcynyszyn LA, Zatzick DF, Chrisman SP, Rivara FP. Child- compared with parent-report ratings on psychosocial measures following a mild traumatic brain injury among youth with persistent post-concussion symptoms. Brain Inj. 2021 Apr 16;35(5):574-586. doi: 10.1080/02699052.2021.1889663. Epub 2021 Mar 18. PMID 33733955
- [Result] McCarty CA, Zatzick DF, Marcynyszyn LA, Wang J, Hilt R, Jinguji T, Quitiquit C, Chrisman SPD, Rivara FP. Effect of Collaborative Care on Persistent Postconcussive Symptoms in Adolescents: A Randomized Clinical Trial. JAMA Netw Open. 2021 Feb 1;4(2):e210207. doi: 10.1001/jamanetworkopen.2021.0207. PMID 33635325
- [Derived] Marcynyszyn LA, McCarty CA, Chrisman SPD, Zatzick DF, Johnson AM, Wang J, Hilt RJ, Rivara FP. Psychometric Properties and Validation of the General Anxiety Disorder 7-Item Scale Among Adolescents With Persistent Post-Concussive Symptoms. Neurotrauma Rep. 2023 Apr 27;4(1):276-283. doi: 10.1089/neur.2022.0075. eCollection 2023. PMID 37139182